CLINICAL TRIAL: NCT01904721
Title: A Safety and Efficacy Study of Bimatoprost in Men With Androgenic Alopecia (AGA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-084
Record Dates: First submitted 2013-07-18; First posted 2013-07-22 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-02

CONDITIONS: Alopecia; Alopecia, Androgenetic; Baldness
MeSH Terms: conditions — Alopecia | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Stage 1: Bimatoprost Solution 1 Twice Daily (Experimental): Stage 1: Bimatoprost Solution 1 applied evenly onto pre-specified area on the scalp twice daily for 28 days.
  Interventions: Drug: Bimatoprost Solution 1
- Stage 1: Bimatoprost Solution 1 Once Daily (Experimental): Stage 1: Bimatoprost Solution 1 applied evenly onto pre-specified area on the scalp once daily for 28 days.
  Interventions: Drug: Bimatoprost Solution 1; Drug: Bimatoprost Vehicle
- Stage 1: Bimatoprost Solution 2 Twice Daily (Experimental): Stage 1: Bimatoprost Solution 2 applied evenly onto pre-specified area on the scalp twice daily for 28 days.
  Interventions: Drug: Bimatoprost Solution 2
- Stage 1: Bimatoprost Solution 2 Once Daily (Experimental): Stage 1: Bimatoprost Solution 2 applied evenly onto pre-specified area on the scalp once daily for 28 days.
  Interventions: Drug: Bimatoprost Solution 2; Drug: Bimatoprost Vehicle
- Stage 2: Bimatoprost Solution 1 Twice Daily (Experimental): Stage 2: Bimatoprost Solution 1 applied evenly onto pre-specified area on the scalp twice daily for 6 months.
  Interventions: Drug: Bimatoprost Solution 1
- Stage 2: Bimatoprost Solution 2 Twice Daily (Experimental): Stage 2: Bimatoprost Solution 2 applied evenly onto pre-specified area on the scalp twice daily for 6 months.
  Interventions: Drug: Bimatoprost Solution 2
- Stage 2: Bimatoprost Vehicle Twice Daily (Placebo Comparator): Stage 2: Bimatoprost Vehicle applied evenly onto pre-specified area on the scalp twice daily for 6 months.
  Interventions: Drug: Bimatoprost Vehicle

INTERVENTIONS:
Drug: Bimatoprost Solution 1 — Bimatoprost Solution 1 applied evenly onto pre-specified area on the scalp daily for 28 days, or daily for 6 months.
  Arms: Stage 1: Bimatoprost Solution 1 Once Daily; Stage 1: Bimatoprost Solution 1 Twice Daily; Stage 2: Bimatoprost Solution 1 Twice Daily
Drug: Bimatoprost Solution 2 — Bimatoprost Solution 2 applied evenly onto pre-specified area on the scalp daily for 28 days, or daily for 6 months.
  Arms: Stage 1: Bimatoprost Solution 2 Once Daily; Stage 1: Bimatoprost Solution 2 Twice Daily; Stage 2: Bimatoprost Solution 2 Twice Daily
Drug: Bimatoprost Vehicle — Bimatoprost Vehicle (placebo) applied evenly onto pre-specified area on the scalp daily for 28 days, or daily for 6 months.
  Arms: Stage 1: Bimatoprost Solution 1 Once Daily; Stage 1: Bimatoprost Solution 2 Once Daily; Stage 2: Bimatoprost Vehicle Twice Daily

SUMMARY:
This is a safety and efficacy study of bimatoprost in male subjects with androgenic alopecia (AGA).

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate male pattern baldness (androgenic alopecia) with ongoing hair loss for at least 1 year
* Willingness to maintain same hair style, length and hair color during study
* Willingness to have micro-dot-tattoo applied to scalp (Stage 2 only)

Exclusion Criteria:

* Drug or alcohol abuse within 12 months
* HIV positive
* Received hair transplants or had scalp reductions
* Use of hair weaves, hair extensions or wigs within 3 months
* Use of minoxidil (oral or topical) and/or low level light treatment "combs" for hair growth within the last 6 months, or expected use during the study
* Application of topical steroids or nonsteroidal anti-inflammatory drugs (NSAIDs) to scalp within 4 weeks

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Fridley, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stage 1: Bimatoprost Solution 1 Twice Daily | Stage 1: Bimatoprost Solution 1 Once Daily | Stage 1: Bimatoprost Solution 2 Twice Daily | Stage 1: Bimatoprost Solution 2 Once Daily | Stage 2: Bimatoprost Solution 1 Twice Daily | Stage 2: Bimatoprost Solution 2 Twice Daily | Stage 2: Bimatoprost Vehicle Twice Daily
Started | 13 | 13 | 12 | 12 | 65 | 65 | 64
Completed | 13 | 13 | 11 | 11 | 57 | 56 | 57
Not Completed | 0 | 0 | 1 | 1 | 8 | 9 | 7
Not completed — Other Reasons | 0 | 0 | 1 | 1 | 2 | 2 | 2
Not completed — Personal Reasons | 0 | 0 | 0 | 0 | 2 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 3 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: Bimatoprost Solution 1 Twice Daily | Stage 1: Bimatoprost Solution 1 Once Daily | Stage 1: Bimatoprost Solution 2 Twice Daily | Stage 1: Bimatoprost Solution 2 Once Daily | Stage 2: Bimatoprost Solution 2 Twice Daily | Stage 2: Bimatoprost Solution 1 Twice Daily | Stage 2: Bimatoprost Vehicle Twice Daily | Total
Number analyzed (Participants) | 13 | 13 | 12 | 12 | 65 | 65 | 64 | 244
Age, Customized [Number; unit: Participants]
  ≥18 to <35 years | 8 | 0 | 3 | 3 | 17 | 18 | 17 | 66
  35 to 49 years | 5 | 13 | 9 | 9 | 48 | 47 | 47 | 178
Sex/Gender, Customized [Number; unit: Participants]
  Male | 13 | 13 | 12 | 12 | 65 | 65 | 64 | 244

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Target Area Hair Count (TAHC)
Description: TAHC was measured using digital imaging analysis and was reported in terminal hairs/centimeters squared (cm^2). A positive change from Baseline indicated improvement (increase in the number of terminal hairs) and a negative change from Baseline indicated worsening (decrease in the number of terminal hairs).
Time Frame: Baseline, Month 6
Population: Modified Intent-to-Treat: all randomized patients in Stage 2 who received study medication and who had both baseline and follow-up TAHC measurements
Measure: Mean (Standard Deviation); unit: terminal hairs/cm2
Arm/Group | Stage 2: Bimatoprost Solution 2 Twice Daily | Stage 2: Bimatoprost Solution 1 Twice Daily | Stage 2: Bimatoprost Vehicle Twice Daily
Number analyzed (Participants) | 63 | 62 | 60
terminal hairs/cm2
  Baseline | 131.3 (55.53) | 140.4 (59.76) | 129.0 (57.42)
  Change from Baseline at Month 6 | 9.3 (23.09) | 12.7 (26.39) | 5.8 (20.95)

2. Primary Outcome: Percentage of Participants in Each Response Category of the Subject Self Assessment in Alopecia (SSA) Score
Description: The SSA score measured scalp hair growth. Using a 7-point scale, participants answered the Question: "Since the start of the study, the amount of my hair has?": Greatly Increased, Moderately Increased, Slightly Increased, Remained the Same, Slightly Decreased, Moderately Decreased or Greatly Decreased. The percentage of participants in each response category is presented.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Stage 2: Bimatoprost Solution 2 Twice Daily | Stage 2: Bimatoprost Solution 1 Twice Daily | Stage 2: Bimatoprost Vehicle Twice Daily
Number analyzed (Participants) | 63 | 62 | 60
Percentage of Participants
  Greatly increased | 4.8 | 6.5 | 0.0
  Moderately increased | 25.4 | 14.5 | 6.7
  Slightly increased | 33.3 | 33.9 | 20.0
  Remained the same | 23.8 | 30.6 | 35.0
  Slightly decreased | 12.7 | 12.9 | 30.0
  Moderately decreased | 0.0 | 1.6 | 6.7
  Greatly decreased | 0.0 | 0.0 | 1.7

3. Secondary Outcome: Percentage of Participants in Each Response Category of the Investigator Global Assessment (IGA) Score
Description: The investigator compared the participant's scalp hair growth at Month 6 to a photograph of the scalp taken at Baseline and using the 7-point IGA score, the investigator answered the question: "Since the start of the study, the amount of the subject's hair has?": Greatly Increased, Moderately Increased, Slightly Increased, Remained the Same, Slightly Decreased, Moderately Decreased or Greatly Decreased. The percentage of participants in each response category is presented.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Stage 2: Bimatoprost Solution 2 Twice Daily | Stage 2: Bimatoprost Solution 1 Twice Daily | Stage 2: Bimatoprost Vehicle Twice Daily
Number analyzed (Participants) | 63 | 62 | 60
Percentage of Participants
  Greatly increased | 4.8 | 11.3 | 0.0
  Moderately increased | 22.2 | 17.7 | 3.3
  Slightly increased | 33.3 | 25.8 | 23.3
  Remained the same | 36.5 | 41.9 | 60.0
  Slightly decreased | 3.2 | 3.2 | 13.3
  Moderately decreased | 0.0 | 0.0 | 0.0
  Greatly decreased | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants in Each Response Category of the Global Panel Review (GPR) Score
Description: At the completion of the study, 3 independent dermatologists using the 7-point GPR score compared photographs of the participant's scalp hair growth at Month 6 to Baseline and answered the question: "Compared with the baseline image, the amount of the subject's hair has?": Greatly Increased, Moderately Increased, Slightly Increased, Remained the Same, Slightly Decreased, Moderately Decreased or Greatly Decreased. The percentage of participants in each response category is presented.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Stage 2: Bimatoprost Solution 2 Twice Daily | Stage 2: Bimatoprost Solution 1 Twice Daily | Stage 2: Bimatoprost Vehicle Twice Daily
Number analyzed (Participants) | 62 | 60 | 58
Percentage of Participants
  Greatly increased | 1.6 | 3.3 | 0.0
  Moderately increased | 9.7 | 15.0 | 0.0
  Slightly increased | 40.3 | 35.0 | 15.5
  Remained the same | 45.2 | 43.3 | 72.4
  Slightly decreased | 3.2 | 3.3 | 10.3
  Moderately decreased | 0.0 | 0.0 | 1.7
  Greatly decreased | 0.0 | 0.0 | 0.0

5. Secondary Outcome: Change From Baseline in Target Area Hair Width (TAHW)
Description: Digital imaging analysis was used to measure TAHW in millimeters/centimeters squared (mm/cm^2). The diameters of all terminal hairs (individual hairs ≥ 30 microns in width) in the target area were summed and reported together. A positive change from Baseline indicated improvement (increase in the diameter of terminal hairs) and a negative change from Baseline indicated worsening (decrease in the diameter of terminal hairs).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/cm2
Arm/Group | Stage 2: Bimatoprost Solution 2 Twice Daily | Stage 2: Bimatoprost Solution 1 Twice Daily | Stage 2: Bimatoprost Vehicle Twice Daily
Number analyzed (Participants) | 63 | 62 | 60
mm/cm2
  Baseline | 7.32 (3.472) | 7.82 (3.764) | 7.30 (3.550)
  Change from Baseline at Month 6 | 0.67 (1.185) | 0.92 (1.435) | 0.05 (1.018)

6. Secondary Outcome: Change From Baseline in Target Area Hair Darkness (TAHD)
Description: Digital imaging analysis was used to measure TAHD. The darkness of all terminal hairs (individual hairs ≥ 30 microns in width) in the target area were summed and divided by total number of terminal hairs in the same target area and was reported as intensity units. A positive change from Baseline indicated improvement (increase in the darkness of terminal hairs) and a negative change from Baseline indicated worsening (decrease in the darkness of terminal hairs).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Intensity Units
Arm/Group | Stage 2: Bimatoprost Solution 2 Twice Daily | Stage 2: Bimatoprost Solution 1 Twice Daily | Stage 2: Bimatoprost Vehicle Twice Daily
Number analyzed (Participants) | 63 | 62 | 60
Intensity Units
  Baseline | 113.77 (19.458) | 115.76 (20.014) | 115.22 (19.879)
  Change from Baseline at Month 6 | -1.63 (17.896) | -6.31 (17.016) | -1.62 (16.763)

ADVERSE EVENTS:
Description: The safety population was defined as all patients who received study medication in the study. The safety population was used to assess adverse events and serious adverse events.
Arm/Group | Stage 1: Bimatoprost Solution 1 Twice Daily | Stage 1: Bimatoprost Solution 1 Once Daily | Stage 1: Bimatoprost Solution 2 Twice Daily | Stage 1: Bimatoprost Solution 2 Once Daily | Stage 2: Bimatoprost Solution 2 Twice Daily | Stage 2: Bimatoprost Solution 1 Twice Daily | Stage 2: Bimatoprost Vehicle Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12 | 0/12 | 1/65 | 2/65 | 0/64
Other Adverse Events (participants affected / at risk) | 5/13 | 4/13 | 7/12 | 1/12 | 25/65 | 25/65 | 7/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Bimatoprost Solution 1 Twice Daily (N=13) | Stage 1: Bimatoprost Solution 1 Once Daily (N=13) | Stage 1: Bimatoprost Solution 2 Twice Daily (N=12) | Stage 1: Bimatoprost Solution 2 Once Daily (N=12) | Stage 2: Bimatoprost Solution 2 Twice Daily (N=65) | Stage 2: Bimatoprost Solution 1 Twice Daily (N=65) | Stage 2: Bimatoprost Vehicle Twice Daily (N=64)
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scapula Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: Bimatoprost Solution 1 Twice Daily (N=13) | Stage 1: Bimatoprost Solution 1 Once Daily (N=13) | Stage 1: Bimatoprost Solution 2 Twice Daily (N=12) | Stage 1: Bimatoprost Solution 2 Once Daily (N=12) | Stage 2: Bimatoprost Solution 2 Twice Daily (N=65) | Stage 2: Bimatoprost Solution 1 Twice Daily (N=65) | Stage 2: Bimatoprost Vehicle Twice Daily (N=64)
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 1
Influenza Like Illness (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Application Site Pruritus (General disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 2 | 1
Electrocardiogram T Wave Amplitude Increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 3 | 1
Growth of Eyelashes (Eye disorders) | 0 | 0 | 0 | 0 | 10 | 0 | 0
Application Site Erythema (General disorders) | 0 | 0 | 0 | 0 | 3 | 5 | 2
Application Site Discoloration (General disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 6 | 2 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 | 6 | 0
Blood Glucose Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Glucose Urine Present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bundle Branch Block Left (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Conjunctival Hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Corneal Irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear Lobe Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.